CLINICAL TRIAL: NCT00870597
Title: Transconjunctival Sutureless 25-Gauge Vitrectomy for Visually Significant Vitreous Floaters in Patients With Multifocal Intraocular Lens
Brief Title: Transconjunctival Sutureless 25-Gauge Vitrectomy
Acronym: TSV-25G
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Oftalmologico de Brasilia (Other)
Collaborators: Federal University of Minas Gerais (Other)
Responsible Party: PATRICK TZELIKIS, UNIVERSIDADE FEDERAL DE MINAS GERAIS
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HOB-03
Record Dates: First submitted 2009-03-26; First posted 2009-03-27 (Estimated); Last update posted 2009-03-27 (Estimated); Status verified 2009-03

CONDITIONS: Visual Acuity
Keywords: Floaters; multifocal IOL; visual complaints; vitrectomy
MeSH Terms: conditions — vitreous floaters | interventions — Vitrectomy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Multifocal IOL implant associated with vitreous opacities that underwent 25-gauge vitrectomy were prospectively analyzed.
  Interventions: Procedure: Multifocal IOL implantation + Vitrectomy
- 2 (Experimental): Multifocal IOL implantation without transconjunctival vitrectomy
  Interventions: Procedure: Multifocal IOL implantation - Vitrectomy

INTERVENTIONS:
Procedure: Multifocal IOL implantation + Vitrectomy — 25-gauge transconjuntival sutureless vitrectomy (TSV)
  Other Names: VITRECTOMY
  Arms: 1
Procedure: Multifocal IOL implantation - Vitrectomy — Multifocal IOL implantation without transconjunctival vitrectomy
  Arms: 2

SUMMARY:
The aim of this study was to evaluate the role of 25-gauge transconjuntival sutureless vitrectomy (TSV) in patients with persistent vitreous floaters who underwent multifocal intraocular lens (IOL) implantation.

DETAILED DESCRIPTION:
Purpose: The aim of this study was to evaluate the role of 25-gauge transconjuntival sutureless vitrectomy (TSV) in patients with persistent vitreous floaters who underwent multifocal intraocular lens (IOL) implantation.

Setting: Hospital Oftalmológico de Brasília, Brasília, DF, Brazil.

Methods: Fourteen eyes of 11 patients with multifocal IOL implant associated with vitreous opacities that underwent 25-gauge vitrectomy were prospectively analyzed. Information collected included near and distance uncorrected visual acuity (UCDVA), best corrected distance visual acuity (BCDVA), and the spherical equivalent (SE) before and 3 months after vitrectomy. Patients were questioned about surgery satisfaction and visual improvement after vitrectomy.

ELIGIBILITY:
Inclusion Criteria:

* disabling vitreous floaters
* Age-related cataract Unsatisfactory correction with glasses

Exclusion Criteria:

* central endothelial cell count less than 2000 cells/mm2
* glaucoma or intraocular pressure greater than 21 mmHg
* amblyopia
* retinal abnormalities
* diabetes mellitus
* steroid or immunosuppressive treatment
* connective tissue diseases

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2007-01; Primary Completion 2008-02 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
The aim of this study was to evaluate the role of 25-gauge transconjuntival sutureless vitrectomy (TSV) in patients with persistent vitreous floaters who underwent multifocal intraocular lens (IOL) implantation | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: PATRICK TZELIKIS, PhD, Principal Investigator — Federal University of Minas Gerais
Locations (1):
- Hospital Oftalmologico de Brasilia, Brasília, Federal District, Brazil